CLINICAL TRIAL: NCT02582190
Title: Colchicine for the Prevention of Atrial Fibrillation Recurrence After Electrical Cardioversion of Persistent Atrial Fibrillation.
Brief Title: COlchicine for the Prevention of Post Electrical Cardioversion Recurrence of AF
Acronym: COPPER-AF
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Investigational Medicinal Product Supplies
Sponsor: Elpen Pharmaceutical Co. Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-IIS-GR-COL
Record Dates: First submitted 2015-10-09; First posted 2015-10-21 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2017-05

CONDITIONS: Atrial Fibrillation
Keywords: electrical cardioversion; persistent atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Colchicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Colchicine group (Other): Colchicine add on therapy in atrial fibrillation
  Interventions: Drug: Colchicine group

INTERVENTIONS:
Drug: Colchicine group — antiarrhythmic therapy plus colchicine & antiarrhythmic therapy alone.
  Other Names: Colchicine in atrial fibrillation

SUMMARY:
There is substantial evidence linking inflammation to the initiation and perpetuation of AF. Although the precise mechanism by which inflammation contributes to the development of AF remains unclear, it has been proposed that inflammation may lead to "atrial myocarditis" with subsequent electrical and structural changes involving both atrial myocytes and extracellular matrix, leading finally to initiation and maintenance of AF. The high incidence of AF in post-operative cardiac surgeries, a state of intense inflammatory process, points out this association. Similarly, in non operative AF, inflammation appears to play a prominent role in both etiology and maintenance of AF. Indeed an increase of inflammatory markers to both paroxysmal and persistent AF was shown by numerous studies.

DETAILED DESCRIPTION:
In particular, CRP levels in patients with persistent AF are higher than in those with paroxysmal AF, and levels in both groups are higher than those in the control group. Moreover, hs-CRP and IL-6 levels have been reported as markers that may identify those patients with a higher risk of AF recurrence after successful electrical cardioversion (EC), providing prognostic information regarding the immediate and long-term success of EC.

CRP is an acute-phase protein and a reliable marker of systemic inflammation. CRP has been shown to specifically bind to phosphatidylcholine on the membranes of myocardial cells which inhibits the exchange of sodium and calcium ions in sarcolemma vesicles, promoting therefore AF development. CRP may also play a part in the structural remodeling; it may induce apoptotic loss of atrial myocytes because of calcium accumulation within atrial myocytes during AF participating also in the clearance of apoptotic atrial myocytes as an opsonin. Myocyte loss is typically accompanied by replacement fibrosis which provides substrate for AF development. IL-6 is one of the most important stimuli of CRP release. As the strongest stimuli of macrophage, TNF-α is in the upstream of this cascade by activating macrophage to release a number of cytokines including IL-6.

Whether inflammatory effects are a consequence of AF or the presence of a pre-existing systemic inflammatory status promotes AF development remains unclear. However, accumulative proofs have implied that both mechanisms may interrelate, suggesting that inflammatory markers are not only a consequence but also a cause.

Consequently, pharmacological interventions with pleiotropic/anti-inflammatory effects might be efficacious in the prevention of AF by modulating inflammatory pathways.(17) Keeping with this, several agents with anti inflammatotory properties as statins, fatty acids, oral glucocorticoids, nonsteroidal anti-inflammatory drugs, angiotensin converting enzyme inhibitors have been administered with controversial results.

Colchicine is a lipid-soluble drug classified as an anti-inflammatory agent. It exerts its anti-inflammatory action without involving the arachidonic acid pathway affected by NSAIDs and glucocorticosteroids. The anti-inflammatory effects of colchicine are attributed to its ability to disrupt the assembly of microtubules in immune-mediated cells. By inhibiting tubulin polymerization, colchicine prevents the activation, degranulation, and migration of neutrophils, which are known initiating factors in inflammatory process. It has also been found to increase leukocyte cyclic adenosine monophosphate levels, inhibit interleukin-1 (IL-1) production by activated neutrophils and down-regulate tumor necrosis factor alpha (TNFa) receptors in macrophages and endothelial cells.

Clinical evidence support that colchicine administration reduced significantly the incidence of AF post-cardiac surgery (POAF) or post-AF ablation and this effect was attributed to the drug anti-inflammatory action. Of note, this effect was accompanied by a significant decrease in inflammatory mediators, IL-6 and CRP as it was shown in post-AF ablation patients.(33) Additional mechanisms may play also a role in the reduction of POAF or post-ablation AF as in vitro or animal studies showed colchicine administration to exert electrophysiological effects related to cytoskeletal disruption.

All patients will undergo echocardiography and blood examination (including thyroid function, renal and liver function tests, lipid assessment, international normalized ratio and foul blood cell count) before EC. Blood samples for CRP, IL-6 and TNFa measurement will be obtained immediately before ECV (day 0), one day after successful ECV (day 1) and after 3 days of colchicine treatment (day 4). Anticoagulation therapy will be instituted according to the current guidelines. If there is indication for transesophageal echocardiography this will be performed prior to EC.

The protocol of electrical cardioversion will be as follows: a shock will be delivered with external paddles positioned in the anterior-apex position connected to an external electrical cardioverter for biphasic external cardioversion. The first shock energy will be delivered at 200 J following a step-up protocol (to 300 J). In case of unsuccessful ECV, a second attempt in anteroposterior position could be made. ECV will be considered successful if sinus rhythm remains 24 hrs after the procedure.

Successfully cardioverted patients will be entered the maintenance phase of the study and treatment will be continued for up to 6 months

ELIGIBILITY:
Inclusion Criteria:

* patients experiencing their first episode of AF of less than 3 months duration will be given no other antiarrhythmic drugs but b-blocker
* In case of recurrent episodes of AF or if AF duration is >3 months patients on antiarrhythmic drugs of class IC or III as first choice.
* men and women
* 18 to 80 years of age
* with persistent AF (sustained for > 7 days) for which electrical cardioversion was indicated.

Exclusion Criteria:

* active inflammatory or infectious disease
* malignancy
* known autoimmune diseases
* corticosteroid or other immunosuppressive or immunomodulatory therapy
* drugs that inhibit CYP3A4 (clarithromycin, azithromycin, ketoconazole, ritonavir, verapamil, and diltiazem)
* moderate or severe hepatic impairment (Child-Pugh class B or C)
* moderate or severe renal failure (≤ 40 ml/min per 1.73 m2)
* acute coronary syndrome within a month before study enrollment
* known blood dyscrasias or gastrointestinal disease
* pregnant and lactating women
* women of childbearing potential not protected by a contraception method -
* patients with atrial flutter will be also excluded unless there is history of coexisting AF.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-12-02 (Estimated); Primary Completion 2018-09-02 (Estimated); Study Completion 2018-09-02 (Estimated)

PRIMARY OUTCOMES:
Number of patients with AF recurrence | 180 days
  Change in AF recurrence from baseline to 180 days

SECONDARY OUTCOMES:
Number of adverse events | 180 days
  Change in adverse events incidence from baseline to 180 days

CONTACTS AND LOCATIONS:
Overall Officials: Nikolaos Fragakis, MD, Principal Investigator — Hippokrateion hospital of Thessaloniki

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Issac TT, Dokainish H, Lakkis NM. Role of inflammation in initiation and perpetuation of atrial fibrillation: a systematic review of the published data. J Am Coll Cardiol. 2007 Nov 20;50(21):2021-8. doi: 10.1016/j.jacc.2007.06.054. Epub 2007 Nov 5. PMID 18021867
- [Background] Aviles RJ, Martin DO, Apperson-Hansen C, Houghtaling PL, Rautaharju P, Kronmal RA, Tracy RP, Van Wagoner DR, Psaty BM, Lauer MS, Chung MK. Inflammation as a risk factor for atrial fibrillation. Circulation. 2003 Dec 16;108(24):3006-10. doi: 10.1161/01.CIR.0000103131.70301.4F. Epub 2003 Nov 17. PMID 14623805
- [Background] Frustaci A, Chimenti C, Bellocci F, Morgante E, Russo MA, Maseri A. Histological substrate of atrial biopsies in patients with lone atrial fibrillation. Circulation. 1997 Aug 19;96(4):1180-4. doi: 10.1161/01.cir.96.4.1180. PMID 9286947
- [Background] Nakamura Y, Nakamura K, Fukushima-Kusano K, Ohta K, Matsubara H, Hamuro T, Yutani C, Ohe T. Tissue factor expression in atrial endothelia associated with nonvalvular atrial fibrillation: possible involvement in intracardiac thrombogenesis. Thromb Res. 2003;111(3):137-42. doi: 10.1016/s0049-3848(03)00405-5. PMID 14678810
- [Background] Bruins P, te Velthuis H, Yazdanbakhsh AP, Jansen PG, van Hardevelt FW, de Beaumont EM, Wildevuur CR, Eijsman L, Trouwborst A, Hack CE. Activation of the complement system during and after cardiopulmonary bypass surgery: postsurgery activation involves C-reactive protein and is associated with postoperative arrhythmia. Circulation. 1997 Nov 18;96(10):3542-8. doi: 10.1161/01.cir.96.10.3542. PMID 9396453
- [Background] Psychari SN, Apostolou TS, Sinos L, Hamodraka E, Liakos G, Kremastinos DT. Relation of elevated C-reactive protein and interleukin-6 levels to left atrial size and duration of episodes in patients with atrial fibrillation. Am J Cardiol. 2005 Mar 15;95(6):764-7. doi: 10.1016/j.amjcard.2004.11.032. PMID 15757607
- [Background] Chung MK, Martin DO, Sprecher D, Wazni O, Kanderian A, Carnes CA, Bauer JA, Tchou PJ, Niebauer MJ, Natale A, Van Wagoner DR. C-reactive protein elevation in patients with atrial arrhythmias: inflammatory mechanisms and persistence of atrial fibrillation. Circulation. 2001 Dec 11;104(24):2886-91. doi: 10.1161/hc4901.101760. PMID 11739301
- [Background] Liu T, Li G, Li L, Korantzopoulos P. Association between C-reactive protein and recurrence of atrial fibrillation after successful electrical cardioversion: a meta-analysis. J Am Coll Cardiol. 2007 Apr 17;49(15):1642-1648. doi: 10.1016/j.jacc.2006.12.042. Epub 2007 Apr 2. PMID 17433956
- [Background] Dernellis J, Panaretou M. Relationship between C-reactive protein concentrations during glucocorticoid therapy and recurrent atrial fibrillation. Eur Heart J. 2004 Jul;25(13):1100-7. doi: 10.1016/j.ehj.2004.04.025. PMID 15231367
- [Background] Conway DS, Buggins P, Hughes E, Lip GY. Predictive value of indexes of inflammation and hypercoagulability on success of cardioversion of persistent atrial fibrillation. Am J Cardiol. 2004 Aug 15;94(4):508-10. doi: 10.1016/j.amjcard.2004.04.070. PMID 15325942
- [Background] Malouf JF, Kanagala R, Al Atawi FO, Rosales AG, Davison DE, Murali NS, Tsang TS, Chandrasekaran K, Ammash NM, Friedman PA, Somers VK. High sensitivity C-reactive protein: a novel predictor for recurrence of atrial fibrillation after successful cardioversion. J Am Coll Cardiol. 2005 Oct 4;46(7):1284-7. doi: 10.1016/j.jacc.2005.06.053. PMID 16198844
- [Background] Wazni O, Martin DO, Marrouche NF, Shaaraoui M, Chung MK, Almahameed S, Schweikert RA, Saliba WI, Natale A. C reactive protein concentration and recurrence of atrial fibrillation after electrical cardioversion. Heart. 2005 Oct;91(10):1303-5. doi: 10.1136/hrt.2004.038661. Epub 2005 May 12. PMID 15890767
- [Background] Loricchio ML, Cianfrocca C, Pasceri V, Bianconi L, Auriti A, Calo L, Lamberti F, Castro A, Pandozi C, Palamara A, Santini M. Relation of C-reactive protein to long-term risk of recurrence of atrial fibrillation after electrical cardioversion. Am J Cardiol. 2007 May 15;99(10):1421-4. doi: 10.1016/j.amjcard.2006.12.074. Epub 2007 Apr 5. PMID 17493472
- [Background] Watanabe E, Arakawa T, Uchiyama T, Kodama I, Hishida H. High-sensitivity C-reactive protein is predictive of successful cardioversion for atrial fibrillation and maintenance of sinus rhythm after conversion. Int J Cardiol. 2006 Apr 14;108(3):346-53. doi: 10.1016/j.ijcard.2005.05.021. Epub 2005 Jun 17. PMID 15964643
- [Background] Korantzopoulos P, Kalantzi K, Siogas K, Goudevenos JA. Long-term prognostic value of baseline C-reactive protein in predicting recurrence of atrial fibrillation after electrical cardioversion. Pacing Clin Electrophysiol. 2008 Oct;31(10):1272-6. doi: 10.1111/j.1540-8159.2008.01177.x. PMID 18811807
- [Background] Smit MD, Maass AH, De Jong AM, Muller Kobold AC, Van Veldhuisen DJ, Van Gelder IC. Role of inflammation in early atrial fibrillation recurrence. Europace. 2012 Jun;14(6):810-7. doi: 10.1093/europace/eur402. Epub 2012 Jan 10. PMID 22237586
- [Background] Van Wagoner DR. Oxidative stress and inflammation in atrial fibrillation: role in pathogenesis and potential as a therapeutic target. J Cardiovasc Pharmacol. 2008 Oct;52(4):306-13. doi: 10.1097/FJC.0b013e31817f9398. PMID 18791466
- [Background] Kallergis EM, Manios EG, Kanoupakis EM, Mavrakis HE, Kolyvaki SG, Lyrarakis GM, Chlouverakis GI, Vardas PE. The role of the post-cardioversion time course of hs-CRP levels in clarifying the relationship between inflammation and persistence of atrial fibrillation. Heart. 2008 Feb;94(2):200-4. doi: 10.1136/hrt.2006.108688. Epub 2007 Jun 17. PMID 17575330
- [Background] Wu N, Xu B, Xiang Y, Wu L, Zhang Y, Ma X, Tong S, Shu M, Song Z, Li Y, Zhong L. Association of inflammatory factors with occurrence and recurrence of atrial fibrillation: a meta-analysis. Int J Cardiol. 2013 Oct 25;169(1):62-72. doi: 10.1016/j.ijcard.2013.08.078. Epub 2013 Sep 8. PMID 24095158
- [Background] Wu J, Corr PB. Influence of long-chain acylcarnitines on voltage-dependent calcium current in adult ventricular myocytes. Am J Physiol. 1992 Aug;263(2 Pt 2):H410-7. doi: 10.1152/ajpheart.1992.263.2.H410. PMID 1510139
- [Background] Nattel S. New ideas about atrial fibrillation 50 years on. Nature. 2002 Jan 10;415(6868):219-26. doi: 10.1038/415219a. PMID 11805846
- [Background] Liu J, Fang PH, Dibs S, Hou Y, Li XF, Zhang S. High-sensitivity C-reactive protein as a predictor of atrial fibrillation recurrence after primary circumferential pulmonary vein isolation. Pacing Clin Electrophysiol. 2011 Apr;34(4):398-406. doi: 10.1111/j.1540-8159.2010.02978.x. Epub 2010 Nov 22. PMID 21091744
- [Background] Rader DJ. Inflammatory markers of coronary risk. N Engl J Med. 2000 Oct 19;343(16):1179-82. doi: 10.1056/NEJM200010193431609. No abstract available. PMID 11036126
- [Background] Cheruku KK, Ghani A, Ahmad F, Pappas P, Silverman PR, Zelinger A, Silver MA. Efficacy of nonsteroidal anti-inflammatory medications for prevention of atrial fibrillation following coronary artery bypass graft surgery. Prev Cardiol. 2004 Winter;7(1):13-8. doi: 10.1111/j.1520-037x.2004.3117.x. PMID 15010623
- [Background] Calo L, Bianconi L, Colivicchi F, Lamberti F, Loricchio ML, de Ruvo E, Meo A, Pandozi C, Staibano M, Santini M. N-3 Fatty acids for the prevention of atrial fibrillation after coronary artery bypass surgery: a randomized, controlled trial. J Am Coll Cardiol. 2005 May 17;45(10):1723-8. doi: 10.1016/j.jacc.2005.02.079. PMID 15893193
- [Background] Young-Xu Y, Jabbour S, Goldberg R, Blatt CM, Graboys T, Bilchik B, Ravid S. Usefulness of statin drugs in protecting against atrial fibrillation in patients with coronary artery disease. Am J Cardiol. 2003 Dec 15;92(12):1379-83. doi: 10.1016/j.amjcard.2003.08.040. PMID 14675569
- [Background] Siu CW, Lau CP, Tse HF. Prevention of atrial fibrillation recurrence by statin therapy in patients with lone atrial fibrillation after successful cardioversion. Am J Cardiol. 2003 Dec 1;92(11):1343-5. doi: 10.1016/j.amjcard.2003.08.023. PMID 14636918
- [Background] Madrid AH, Bueno MG, Rebollo JM, Marin I, Pena G, Bernal E, Rodriguez A, Cano L, Cano JM, Cabeza P, Moro C. Use of irbesartan to maintain sinus rhythm in patients with long-lasting persistent atrial fibrillation: a prospective and randomized study. Circulation. 2002 Jul 16;106(3):331-6. doi: 10.1161/01.cir.0000022665.18619.83. PMID 12119249
- [Background] Tveit A, Seljeflot I, Grundvold I, Abdelnoor M, Smith P, Arnesen H. Effect of candesartan and various inflammatory markers on maintenance of sinus rhythm after electrical cardioversion for atrial fibrillation. Am J Cardiol. 2007 Jun 1;99(11):1544-8. doi: 10.1016/j.amjcard.2007.01.030. Epub 2007 Apr 16. PMID 17531578
- [Background] Ferron GM, Rochdi M, Jusko WJ, Scherrmann JM. Oral absorption characteristics and pharmacokinetics of colchicine in healthy volunteers after single and multiple doses. J Clin Pharmacol. 1996 Oct;36(10):874-83. doi: 10.1002/j.1552-4604.1996.tb04753.x. PMID 8930773
- [Background] Terkeltaub RA. Colchicine update: 2008. Semin Arthritis Rheum. 2009 Jun;38(6):411-9. doi: 10.1016/j.semarthrit.2008.08.006. Epub 2008 Oct 29. PMID 18973929
- [Background] Van Wagoner DR. Colchicine for the prevention of postoperative atrial fibrillation: a new indication for a very old drug? Circulation. 2011 Nov 22;124(21):2281-2. doi: 10.1161/CIRCULATIONAHA.111.057075. No abstract available. PMID 22105193
- [Background] Deftereos S, Giannopoulos G, Kossyvakis C, Efremidis M, Panagopoulou V, Kaoukis A, Raisakis K, Bouras G, Angelidis C, Theodorakis A, Driva M, Doudoumis K, Pyrgakis V, Stefanadis C. Colchicine for prevention of early atrial fibrillation recurrence after pulmonary vein isolation: a randomized controlled study. J Am Coll Cardiol. 2012 Oct 30;60(18):1790-6. doi: 10.1016/j.jacc.2012.07.031. Epub 2012 Oct 3. PMID 23040570
- [Background] Kamkin A, Kiseleva I, Wagner KD, Scholz H, Theres H, Kazanski V, Lozinsky I, Gunther J, Isenberg G. Mechanically induced potentials in rat atrial fibroblasts depend on actin and tubulin polymerisation. Pflugers Arch. 2001 Jul;442(4):487-97. doi: 10.1007/s004240100564. PMID 11510879
- [Background] Climent V, Marin F, Mainar L, Roldan V, Garcia A, Martinez JG, Lip GY. Influence of electrical cardioversion on inflammation and indexes of structural remodeling, in persistent atrial fibrillation. Int J Cardiol. 2009 Feb 20;132(2):227-32. doi: 10.1016/j.ijcard.2007.11.044. Epub 2008 Jan 30. PMID 18234374
- [Background] Nichol G, McAlister F, Pham B, Laupacis A, Shea B, Green M, Tang A, Wells G. Meta-analysis of randomised controlled trials of the effectiveness of antiarrhythmic agents at promoting sinus rhythm in patients with atrial fibrillation. Heart. 2002 Jun;87(6):535-43. doi: 10.1136/heart.87.6.535. PMID 12010934